CLINICAL TRIAL: NCT06736613
Title: Cerebral Spinal Fluid Circulating Tumor DNA (ctDNA) Analysis in Patients With Aggressive B-cell Lymphoma Receiving Front Line Therapy and at High Risk for Central Nervous System Relapse
Brief Title: A Study of Circulating Tumor DNA (ctDNA) Testing for People With B-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-336
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Stage III High Grade B-Cell Lymphoma; Stage IV High Grade B-Cell Lymphoma; DLBCL - Diffuse Large B Cell Lymphoma; Intravascular Large B-Cell Lymphoma; Diffuse Large B Cell Lymphoma of Breast; Diffuse Large B Cell Lymphoma of Testis; HIV-associated Diffuse Large B Cell Lymphoma; Double Expressor DLBCL
Keywords: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Stage III High Grade B-Cell Lymphoma; Stage IV High Grade B-Cell Lymphoma; DLBCL - Diffuse Large B Cell Lymphoma; Intravascular Large B-Cell Lymphoma; Diffuse Large B Cell Lymphoma of Breast; Diffuse Large B Cell Lymphoma of Testis; HIV-associated Diffuse Large B Cell Lymphoma; Double expressor DLBCL; Circulating Tumor DNA; ctDNA; Memorial Sloan Kettering Cancer Center; 24-336
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Diffuse large B-cell lymphoma (DLBCL) i (Experimental): Participants will be deemed clinically high-risk for CNS relapse. Participants will be considered to be high-risk for CNS relapse as determined by CNS-IPI score, pathological characteristics such as the presence of MYC, BCL2 and/or BCL6 translocations and specific extranodal involvement such as breast, renal, adrenal, nasopharyngeal, epidural/paraspinal involvement
  Interventions: Diagnostic Test: Cerebral Spinal Fluid ctDNA

INTERVENTIONS:
Diagnostic Test: Cerebral Spinal Fluid ctDNA — MSK's Diagnostic Molecular Pathology core has developed and validated a CSF ctDNA assay which has been approved by New York State Department of Health as of 2019

SUMMARY:
The purpose of this study is to find out how many people with B-cell lymphoma who are at high risk for central nervous system/CNS relapse test positive for cerebral spinal fluid/CSF ctDNA but test negative for CNS involvement using standard tests. The study will also look at how often CNS relapse happens in people with and without detected CSF ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent.
* Ability and willingness to comply with the requirements of the study protocol.
* Age ≥ 18 years old.
* Diagnosis of the following histologies according to the 2016 WHO Classification for Mature Lymphoid Neoplasms81 along with a specific high-risk criteria for CNS relapse if indicated as certain diagnoses in of themselves are high-risk alone:

  1. Diffuse Large B-cell Lymphoma (DLBCL) with CNS IPI score ≥ 4.
  2. Stage III/IV High Grade B-cell lymphoma (HGBCL) with MYC, BCL2, and/or BCL6 translocations
  3. Primary DLBCL of Breast
  4. Primary DLBCL of Testis
  5. Primary Cutaneous DLBCL, Leg Type
  6. Intravascular Large B-cell Lymphoma
  7. Stage III/IV HIV-associated DLBCL
  8. Double expressor DLBCL (co-expression of MYC ≥ 40% and BCL2 ≥ 50% without translocations) with a CNS IPI score ≥ 3
  9. DLBCL with the following extranodal involvement AND CNS IPI score ≥ 3:

  i. Adrenal ii. Breast iii. Bone Marrow with pathological overt morphological involvement iv. Epidural/Paraspinal v. Nasal/parasinus with local invasion such as bone destruction vi. Renal viii. Uterine ix. Testis xi. Skull involvement without direct invasion into CNS/brain parenchyma
* Transformed DLBCL from any indolent B-cell lymphoma is permitted (as long as there is no prior history of CNS involvement).
* Planned to receive standard chemoimmunotherapy.
* Patient is able to undergo lumbar puncture without any contraindications which include but are not limited to altered mental status, increased intracranial pressure due to any CNS lesion (mass, abscess), overlying skin infection at the site of LP, inability to safely access CSF due to lymphomatous involvement (i.e. epidural mass), or inability to hold antiplatelet or anticoagulation safely for the procedure to be performed.
* No systemic therapy prior to study enrollment for an aggressive B-cell lymphoma is permitted. Treatment for a history of indolent lymphoma is permitted. Systemic corticosteroids are permitted (must be ≤7 days and tapered down to prednisone ≤ 20 mg oral/day or steroid equivalent by first day of anthracycline treatment). Clinical exceptions in regards to steroid management can be made after discussion with PI.
* ECOG performance status of 0 to 2.

Exclusion Criteria:

* Active systemic therapy for another malignancy (other than indolent B-cell lymphoma) within 2 years; local/regional therapy with curative intent such as surgical resection or localized radiation within 2 years of treatment is permitted.
* Active concurrent malignancy with the exception of basal cell or localized squamous cell skin carcinoma, localized prostate cancer, or other localized carcinomas such as carcinoma in situ of cervix, breast, or bladder.
* Any uncontrolled illness that in the opinion of the investigator would preclude administration of curative intent chemoimmunotherapy (e.g. significant active infections, hypertension, angina, arrhythmias, pulmonary disease, or autoimmune dysfunction).
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 2 weeks prior to Cycle 1, Day 1.
* Psychiatric illness or social situations that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-12-11 (Estimated); Study Completion 2027-12-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of positive cerebral spinal fluid/CSF ctDNA | up to 2 years
  The primary objective is to describe the incidence of positive CSF ctDNA in participants at high-risk for CNS relapse

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lue, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org